CLINICAL TRIAL: NCT04789005
Title: Comparison of Intravenous Phenylephrine and Norepinephrine for Treatment of Spinal-induced Hypotension in Caesarian Deliveries
Brief Title: Comparison of Phenylephrine and Norepinephrine for Spinal-induced Hypotension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, ALLEN SUWAL, Resident Anaesthesiology, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 439/(6-11)E²/076/077
Record Dates: First submitted 2021-02-10; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Spinal Induced-hypotension
MeSH Terms: interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phenylephrine group (Active Comparator): Phenylephrine 100mcg was administered manually by the anaesthesiologist every time the SBP was 20% lower than baseline and the HR ≥60 bpm.
  Interventions: Drug: Phenylephrine
- Norepinephrine group (Experimental): Norepinephrine 8mcg was administered manually by the anaesthesiologist every time the SBP was 20% lower than baseline and the HR ≥60 bpm.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine 8mcg was administered manually by the anaesthesiologist every time the SBP was 20% lower than baseline and the HR ≥60 bpm.
  Other Names: Norepinephrine group
  Arms: Norepinephrine group
Drug: Phenylephrine — Phenylephrine 100mcg was administered manually by the anaesthesiologist every time the SBP was 20% lower than baseline and the HR ≥60 bpm.
  Other Names: Phenylepherine group
  Arms: Phenylephrine group

SUMMARY:
Hypotension after spinal anaesthesia for cesarean deliveries is frequently encountered. Phenylephrine an α-agonist is commonly used for the prevention and treatment of spinal-induced hypotension. Phenylephrine causes baroreceptor-mediated bradycardia leading to subsequent reduction in cardiac output. Preservation of heart rate and cardiac output is important in high-risk conditions such as placental insufficiency, fetal distress and maternal cardiac disease. Recently, norepinephrine has been found as effective as phenylephrine in treatment of spinal induced hypotension. When norepinephrine is used as a bolus, it is effective at maintaining blood pressure while also conferring a greater heart rate and cardiac output compared to phenylephrine.

ELIGIBILITY:
Inclusion Criteria:

Elective cesarean delivery under spinal anaesthesia ASA PS II Age ≥18 years Singleton pregnancy beyond 37 weeks' gestation Weight between 50 and 100 kg Height between 150 and 180 cm

Exclusion Criteria:

Patient refusal to participate Allergy or hypersensitivity to Norepinephrine or Phenylephrine Preexisting or pregnancy-induced hypertension Cardiovascular or cerebrovascular disease Fetal abnormalities Use of monoamine oxidase inhibitors or tricyclic antidepressants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
To compare blood pressure between two groups. | 6 months
To compare percentage of incidence of hypotension between two groups. | 6 months
compare percentage of incidence of bradycardia between the two groups | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Tribhuvan university teaching hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No